CLINICAL TRIAL: NCT01144598
Title: Time to DMARD Treatment and Actual Work Limitation of Patients With Rheumatoid Arthritis in Turkey
Brief Title: Time to DMARD (Disease-Modifying Anti-Rheumatic Drug) Treatment and Actual Work Limitation of Patients With Rheumatoid Arthritis in Turkey
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P12-087
Record Dates: First submitted 2010-05-28; First posted 2010-06-15 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Disease-Modifying Anti-Rheumatic Drug; Work Limitation
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Turkish patients with rheumatoid arthritis

SUMMARY:
The objective is to measure time delay from onset of symptoms to diagnosis and time to disease-modifying anti-rheumatic drug treatments in Turkish patients with rheumatoid arthritis. The investigators will also evaluate actual work limitation status of patients and impact of demographic and clinical factors on work limitations in rheumatoid arthritis patients.

DETAILED DESCRIPTION:
This post marketing observational study will be conducted in cross-sectional, non-interventional, multi-center format in Turkey. As this is a post marketing observational study, Abbott is not involved in the product supply since the drug is being used according to the approved marketing label and is to be prescribed by the physician under usual and customary practice of physician prescription.

Subjects will be recruited from rheumatology outpatient clinics of university hospitals and/or private offices.

Patients diagnosed with rheumatoid arthritis who had received at least one disease-modifying anti-rheumatic drug, who are already employed at a paid work and able to provide disease history data will be included.

Patient data will be collected with a single visit. During the single visit, all required demographic and clinical data will be recorded on the case report forms by the investigators and every subject will be asked to fill out the Work Productivity and Activity Impairment questionnaire and the Health Assessment Questionnaire - Disability Index.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis by a specialist or by the treating rheumatologist
* Treated with at least one disease-modifying anti-rheumatic drug or biologics
* Patients over 18 years
* Patients already employed at a paid work
* Patients able to provide data for disease history
* Able to provide written consent to release information for this study

Exclusion Criteria:

* Patients who cannot provide necessary outcome measurements for any reason will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As this study is non-randomized, the normal study population and design requirements for power calculations are not met. Therefore, the results of the following should be interpreted as indicative only. Subjects will be recruited from rheumatology outpatient clinics of university hospitals and/or private offices.
  Patients diagnosed with rheumatoid arthritis who had received at least one disease-modifying anti-rheumatic drug, who are already employed at a paid work and are able to provide disease history data will be included.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Gucuk, MD, Study Director — Abbott
Locations (21):
- Turkey (Türkiye) (21):
  - Site Reference ID/Investigator# 39111, Adana
  - Site Reference ID/Investigator# 39102, Ankara
  - Site Reference ID/Investigator# 39104, Ankara
  - Site Reference ID/Investigator# 39109, Ankara
  - Site Reference ID/Investigator# 52448, Ankara
  - Site Ref # / Investigator 52451, Antalya
  - Site Reference ID/Investigator# 52442, Aydin
  - Site Reference ID/Investigator# 52447, Bursa
  - Site Reference ID/Investigator# 52446, Bursa
  - Site Ref # / Investigator 52443, Denizli
  - Site Reference ID/Investigator# 52444, Denizli
  - Site Reference ID/Investigator# 52449, Gaziantep
  - Site Reference ID/Investigator# 52450, Gaziantep
  - Site Reference ID/Investigator# 39107, Istanbul
  - Site Reference ID/Investigator# 39106, Istanbul
  - Site Reference ID/Investigator# 39103, Istanbul
  - Site Reference ID/Investigator# 39108, Izmir
  - Site Reference ID/Investigator# 36442, Izmir
  - Site # / Investigator 59224, Izmir
  - Site Ref # / Investigator 59225, Izmir
  - Site Ref # / Investigator 59226, Izmir

RESULTS

PARTICIPANT FLOW:
Groups:
- Turkish Patients With Rheumatoid Arthritis: Patients diagnosed with rheumatoid arthritis who had received at least one disease-modifying anti-rheumatic drug, who are already employed at a paid work and able to provide disease history data.
Period: Overall Study
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Started | 356
Analysis Population | 356
Completed | 356
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 356
Age, Customized [Number; unit: participants]
  Less than 30 years | 49
  30 to 40 years | 122
  41 to 50 years | 120
  51 to 60 years | 53
  Over 60 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216
  Male | 140

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Disease Duration: Time From Diagnosis to Disease-Modifying Anti-Rheumatic Drug Treatment in Rheumatoid Arthritis
Description: The time elapsed from diagnosis of rheumatoid arthritis to initiation of treatment with disease-modifying anti-rheumatic drugs (DMARDs).
Time Frame: Day 1
Population: All participants with available information were included in the analysis.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 355
Months | 11.7177 (22.513)

2. Secondary Outcome: Work Limitation: Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: The HAQ-DI measures physical function by assessing the ability to perform daily living tasks. Each task is rated from 0 (no difficulty) to 3 (unable to do). The total score ranges from 0 to 3. Higher scores indicate impairment.
Time Frame: Day 1
Population: All participants who completed the rating scales were included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 356
Units on a scale | 0.96 (0.7)

3. Secondary Outcome: Work Limitation: Work Productivity and Activity Impairment (WPAI) Questionnaire
Description: The WPAI evaluates the ability to work and perform regular activities. The scale yields 4 types of scores (range 0 to 100): Absenteeism (work time missed); Presenteeism (impairment at work/reduced on-the-job effectiveness); Work Productivity Loss (overall work impairment/absenteeism plus presenteeism); and Activity Impairment. Higher scores indicate impairment.
Time Frame: Day 1
Population: All participants who completed the rating scales were included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 356
Units on a scale
  WPAI (Absenteeism) | 12.3 (25.2)
  WPAI (Presenteeism) | 39.1 (29.2)
  WPAI (Work Productivity Loss) | 42.3 (32.2)
  WPAI (Activity Impairment) | 38.7 (27.9)

4. Secondary Outcome: Evaluation of Global Rheumatoid Arthritis Severity Scale
Description: Global rheumatoid arthritis severity was assessed by asking the participants to consider all the ways their rheumatoid arthritis affected them and to rate how they were doing on a scale of 0 (very well) to 10 (very poor).
Time Frame: Day 1
Population: All participants with available information were included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 356
Units on a scale | 4.07 (2.50)

5. Secondary Outcome: Evaluation of Disease Activity Score 28 (DAS28)
Description: The DAS28 index measures disease activity in rheumatoid arthritis and is derived from the number of swollen/tender joints, laboratory tests of inflammation, and participant assessment of global health (by marking a 100 mm line from "very good" to "very bad"). A higher score indicates worse control of disease. A DAS28 less than 3.2 indicates low disease activity and a DAS28 greater than 5.1 indicates high disease activity.
Time Frame: Day 1
Population: All participants with available information were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 353
Participants
  DAS28 less than 2.6 | 84
  DAS28 2.6 to less than 3.2 | 64
  DAS28 3.2 to less than or equal to 5.1 | 129
  DAS28 greater than 5.1 | 76

6. Secondary Outcome: Evaluation of Visual Analog Scale (VAS) for Pain and Fatigue
Description: Participants rated their pain and fatigue using a visual analog scale from 0 to 10, where 10 was the worst case.
Time Frame: Day 1
Population: Participants who provided a visual analog scale rating for pain and fatigue were included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 355
Units on a scale | 4.24 (2.77)

7. Secondary Outcome: Number of Disease Modifying Anti-Rheumatic Drugs
Description: The number of disease-modifying anti-rheumatic drugs (DMARDs) that participants were taking to treat their rheumatoid arthritis.
Time Frame: Day 1
Population: All participants with available information were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 356
Participants
  Taking 1 DMARD | 44
  Taking 2 DMARDs | 94
  Taking 3 DMARDs | 78
  Taking more than 3 DMARDs | 35

8. Secondary Outcome: Biologics Usage
Description: Biologic treatments participants were taking for their rheumatoid arthritis.
Time Frame: Day 1
Population: All participants with available information were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 356
Participants
  Taking 1 biologic plus 1 DMARD | 85
  Taking 2 biologics plus 1 DMARD | 16
  Taking more than 2 biologics plus 1 DMARD | 4

9. Secondary Outcome: Stiffness Duration
Description: Participants' duration of morning joint stiffness.
Time Frame: Day 1
Population: All participants with available information were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 355
Participants
  0 to 10 minutes | 161
  11 to 30 minutes | 78
  31 to 60 minutes | 54
  61 minutes or longer | 62

10. Secondary Outcome: Number of Comorbidities
Description: Number of comorbid (coexisting) medical conditions of the study participants.
Time Frame: Day 1
Population: All participants with available information were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 356
Participants
  No comorbid conditions | 259
  One comorbid condition | 72
  Two comorbid conditions | 22
  Three or more comorbid conditions | 3

11. Secondary Outcome: Rheumatoid Factor
Description: Rheumatoid factor test results.
Time Frame: Day 1
Population: All participants with available information were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 344
Participants
  Rheumatoid factor positive | 248
  Rheumatoid factor negative | 96

12. Secondary Outcome: Anti-cyclic Citrullinated Peptide
Description: Anti-cyclic citrullinated peptide (anti-CCP) test results.
Time Frame: Day 1
Population: All participants with available information were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 256
Participants
  Anti-CCP positive | 181
  Anti-CCP negative | 75

13. Secondary Outcome: Sedimentation Rate
Description: The erythrocyte (red blood cell) sedimentation rates of study participants were assessed.
Time Frame: Day 1
Population: All participants with available information were included in the analysis.
Measure: Mean (Standard Deviation); unit: millimeters/hour
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 350
millimeters/hour | 27.53 (21.67)

14. Secondary Outcome: Number of Deformities at Inspection
Description: The number of joint deformities of the study participants.
Time Frame: Day 1
Population: All participants with available information were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 354
Participants
  No deformities | 221
  One deformity | 34
  Two deformities | 33
  Three or more deformities | 66

15. Secondary Outcome: Evaluation of Rheumatoid Arthritis Treatments Duration
Description: Time elapsed from onset of symptoms to diagnosis of rheumatoid arthritis (that is, from the first rheumatoid arthritis-related symptoms to diagnosis by a related specialist) and the time elapsed from diagnosis with rheumatoid arthritis to initiation of anti-tumor necrosis factor (anti-TNF) treatment.
Time Frame: Day 1
Population: All participants with available information were included in the analysis.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Number analyzed (Participants) | 355
Months
  Time from symptoms to diagnosis (n=355) | 16.2468 (28.680)
  Time from diagnosis to anti-TNF treatment (n=104) | 68.57 (90.22)

ADVERSE EVENTS:
Time Frame: Participants were interviewed during a single visit. Adverse events which were observed/reported during this single visit were to be subject to local pharmacovigilance requirements, however, no adverse event or serious adverse event reports were made.
Arm/Group | Turkish Patients With Rheumatoid Arthritis
Serious Adverse Events (participants affected / at risk) | 0/356
Other Adverse Events (participants affected / at risk) | 0/356

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.